CLINICAL TRIAL: NCT04998448
Title: History of Exposure to Endocrine Disruptors in Women With Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO21065
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Polycystic Ovary Syndrome; Exposure to Endocrine Disruptors
Keywords: Polycystic ovary syndrome; Endocrine disruptors
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: women aged 18 to 50 years, premenopausal, with polycystic ovary syndrome
- Controls: women aged 18 to 50 years, premenopausal, without polycystic ovary syndrome.

SUMMARY:
Polycystic ovary syndrome is a common endocrine disorder that affects between 7% and 14% of women of childbearing age, leading to impaired fertility, clinical and biological hyperandrogenism.

Long-term complications such as metabolic disorders, cardiovascular disease and hormone-dependent cancers make it a major public health problem.

The physiopathology of this syndrome is complicated and still poorly understood, probably multifactorial origin, resulting from the interaction between many factors (genetics, lifestyle, environment).

The environment has also an important role in the development of polycystic ovary syndrome : diet, exposure to pollutants and endocrine disruptors.

There are many sources of exposure to environmental toxins and it is essential to better understand their impact on our health.

Our study aims to assess the association between exposure to endocrine disruptors and development of polycystic ovary syndrome.

The population involved in the study includes patients aged 18 to 50 years, premenopausal, consulting in the gynecology department of the university hospital of Reims.

The "cases" patients will be patients with polycystic ovary syndrome. The "controls" patients will be patients without polycystic ovary syndrome. Statistical analysis will determine whether "cases" are more exposed to endocrine disruptors than "controls".

DETAILED DESCRIPTION:
Polycystic ovary syndrome is a common endocrine disorder that affects between 7% and 14% of women of childbearing age, leading to impaired fertility, clinical and biological hyperandrogenism.

Long-term complications such as metabolic disorders, cardiovascular disease and hormone-dependent cancers make it a major public health problem.

The physiopathology of this syndrome is complicated and still poorly understood, probably multifactorial origin, resulting from the interaction between many factors (genetics, lifestyle, environment).

The environment has also an important role in the development of polycystic ovary syndrome : diet, exposure to pollutants and endocrine disruptors.

There are many sources of exposure to environmental toxins and it is essential to better understand their impact on our health.

Our study aims to assess the association between exposure to endocrine disruptors and development of polycystic ovary syndrome.

The population involved in the study includes patients aged 18 to 50 years, premenopausal, consulting in the gynecology department of the university hospital of Reims.

The "cases" patients will be patients with polycystic ovary syndrome. The "controls" patients will be patients without polycystic ovary syndrome. Statistical analysis will determine wether "cases" are more exposed to endocrine disruptors than "controls". "Cases" and "controls" will be matched on age (+/- 5 years).

The statistical analysis consists of description of data (mean and standard deviation, number and percentage) and comparison of exposure to toxicants and endocrine disruptors according to the "cases" and "controls" group by univariate analysis (tests of Student, Wilcoxon, Chi 2 or Fisher's exact) then multivariate (logistic regression).

ELIGIBILITY:
inclusion criteria for "cases" :

* age 18 to 50 years
* premenopausal
* diagnostic of PCOS has been made according to Rotterdam criteria
* followed in the gynecology and endocrinology departments at the university hospital of Reims.
* agreeing to participate in the study

inclusion criteria for "controls"

* age 18 to 50 years
* premenopausal
* diagnostic of PCOS can be excluded du to the absence of menstrual cycle disorders and absence of clinical signs of hyperandrogenism
* followed in the gynecology and endocrinology departments at the university hospital of Reims.
* agreeing to participate in the study

exclusion criteria:

* under the of 18 years or over 50 years
* menopausal
* refusing to participate in the study
* protected by law

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population involved in the study includes patients aged 18 to 50 years, premenopausal, consulting in the gynecology department of the university hospital of Reims The "cases" patients will be patients with polycystic ovary syndrome. The "controls" patients will be patients without polycystic ovary syndrome. "Cases" and "controls" will be matched on age (+/- 5 years).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Survey form on exposure to endocrine disruptors | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France